CLINICAL TRIAL: NCT06216925
Title: Teen Mom Study: A Confirmatory Pragmatic Cluster Randomized Controlled Trial
Brief Title: Teen Mom Study: A Confirmatory Pragmatic Cluster RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: University of Alabama at Birmingham (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Abigail Gamble, Associate Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-409; P50MD017338 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Behavior; Physical Activity; Gestational Weight Gain; Arterial Pressure
Keywords: Pregnancy; Adolescent; Mobile Health
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- #BabyLetsMove (Experimental): For 24 weeks, participants will wear a Fitbit activity tracker (continually) and receive interactive self-monitoring and tailored feedback text messages (twice per week), tailored skills training texts and materials (once per week), and peer health coaching (once every other week). In addition, the participants will receive ancillary healthy food to allay food insecurity, nutritional counseling, and clinical care referrals once every three months.
  Interventions: Behavioral: #BabyLetsMove
- WIC Antenatal Care (Active Comparator): The participants will receive ancillary healthy food to allay food insecurity, nutritional counseling, and clinical care referrals once every three months.
  Interventions: Behavioral: WIC Antenatal Care

INTERVENTIONS:
Behavioral: #BabyLetsMove — Description of #BabyLetsMove
  Arms: #BabyLetsMove
Behavioral: WIC Antenatal Care — Description
  Arms: WIC Antenatal Care

SUMMARY:
The goal of this clinical trial is to test the effectiveness of #BabyLetsMove - a 24-week mobile Health and peer health coaching intervention paired with the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) - to increase physical activity and reduce sedentary behavior in pregnant, Black teens in the Mississippi Delta. The main questions it aims to answer are:

* Does #BabyLetsMove increase objective moderate-to-vigorous physical activity and decrease sedentary behavior from ≤16 to 26- and 36-gestational weeks compared to usual WIC care alone?
* Does # BabyLetsMove decrease the rate of gestational weight gain and mean arterial pressure from ≤16 to 26- and 36-gestational weeks compared to usual WIC care alone?
* Is #BabyLetsMove a feasible and acceptable intervention according to the RE-AIM framework?
* Using the Practical, Robust Implementation and Sustainability Model and the Consolidated Framework for Implementation Research, what are the barriers to organizational uptake and how can strategies be improved for future testing?

Participants will be given three empirically supported behavior goals including (1) watching ≤2 hours of TV or other screen time per day, and (2) walking ≥10,000 steps per day - or - (3) engaging in ≥20 minutes of organized exercise per day.

Researchers will compare the #BabyLetsMove groups to the WIC care only groups to see if the #BabyLetsMove intervention improves traditional WIC care for bettering health outcomes ( amongst pregnant, Black teens in the Mississippi Delta.

DETAILED DESCRIPTION:
The "Teen Mom Study: A Hybrid Cluster Randomized Trial" proposes a pragmatic, multilevel, type I study design to test the effectiveness of #BabyLetsMove - a 24-week mHealth and peer health coaching intervention paired with the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) - to increase physical activity and reduce sedentary behavior in pregnant, Black teens in the Mississippi Delta. Concurrently, a robust implementation evaluation will be conducted to determine feasibility and acceptability and to identify threats to organizational uptake, scalability, and sustainability. The intervention will be delivered remotely in partnership with WIC (Mississippi State Department of Health), the Telehealth Center of Excellence, and Myrlie Evers-Williams Institute (University of Mississippi Medical Center). The intervention is based on formative data from the "Teen Mom Study" and uses a theory-based, multi-level systems change approach. At the systems level, racially concordant young adult (18 to 25 years) WIC moms (n=4) are undergoing paid skills training in evidence-based peer health coaching to first, address social needs in pregnant teens and second, provide support for self-directed behavior change. At the individual level, pregnant, Black teens will be given three empirically supported behavior goals including (1) watching ≤2 hours of TV or other screen time per day, and (2) walking ≥10,000 steps per day - or - (3) engaging in ≥20 minutes of organized exercise per day. The intervention is designed to build social cognition, affect, and skills using four intervention components - a wearable tracker, interactive self-monitoring text messages with automated feedback, tailored skills training texts linked to digital materials, and peer health coaching. The central hypothesis is that augmenting usual WIC care with #BabyLetsMove will improve WIC's capacity to serve rural families and empower pregnant, Black teens to prioritize and improve their health. The primary aim is to determine the effect of #BabyLetsMove compared to usual WIC care on objective moderate-to-vigorous physical activity and sedentary behavior from ≤16 to 26- and 36-gestational weeks using a parallel cluster randomized trial. Secondary aim 1 will use wearables plus remote monitoring to measure and explore patterns of gestational weight gain and mean arterial pressure within/across conditions. Secondary aim 2.a. will use the RE-AIM framework to evaluate the feasibility and acceptability of #BabyLetsMove, and Secondary aim 2.b. will use the Practical, Robust Implementation and Sustainability Model and the Consolidated Framework for Implementation Research to identify threats to organizational uptake and to develop implementation strategies for future testing. This is believed to be the first digital health intervention study designed with/for a pregnant adolescent population. This study will add to our understanding of optimal mHealth and peer health coaching interventions; advance implementation science literature by studying a scalable and sustainable intervention in a novel setting; and contribute to the urgent national agenda to advance Black maternal health equity.

ELIGIBILITY:
Inclusion Criteria:

* Less than 16 weeks pregnant
* Black or African-American
* Between 15 and 19 years of age (inclusive)
* Enrolled in WIC
* Residing in 1 of 12 counties constituting the Mississippi Delta region
* Singleton pregnancy
* Planning to carry the fetus to term
* English speaking
* Possession of a mobile device

Exclusion Criteria:

* Individuals with physical activity restrictions

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Moderate-to-Vigorous Physical Activity at 26 Weeks Gestation | Baseline to 26 weeks gestation
  Actigraph accelerometry (GT9X Link) will be used to measure MVPA (>3 METs) and SB (<1.5 METs) for 24 hours per day, over a 7-day period,155 across 3-time points (Table 5). Accelerometers will be worn on teens' non-dominant wrists to record raw acceleration data using a sampling rate of 100 Hz and converted into objective measures.
Change in Moderate-to-Vigorous Physical Activity at 36 Weeks Gestation | Baseline to 36 weeks gestation
  Actigraph accelerometry (GT9X Link) will be used to measure MVPA (>3 METs) for 24 hours per day, over a 7-day period. Accelerometers will be worn on teens' non-dominant wrists to record raw acceleration data using a sampling rate of 100 Hz and converted into objective measures.
Change in Sedentary Behavior at 26 Weeks Gestation | Baseline to 26 weeks gestation
  Actigraph accelerometry (GT9X Link) will be used to measure sedentary behavior (<1.5 METs) for 24 hours per day, over a 7-day period. Accelerometers will be worn on teens' non-dominant wrists to record raw acceleration data using a sampling rate of 100 Hz and converted into objective measures.
Change in Sedentary Behavior at 36 Weeks Gestation | Baseline to 36 weeks gestation
  Actigraph accelerometry (GT9X Link) will be used to measure sedentary behavior (<1.5 METs) for 24 hours per day, over a 7-day period. Accelerometers will be worn on teens' non-dominant wrists to record raw acceleration data using a sampling rate of 100 Hz and converted into objective measures.

SECONDARY OUTCOMES:
Change in Gestational Weight Gain at 26 Weeks Gestation | Baseline to 26 weeks gestation
  Body weight will be measured at each time point using Tanita MC-780U scale to assess gestational weight gain (GWG). Participants will use a BodyTrace scale linked to a secure monitoring system for weekly self-weighing monitored by health coaches. If weight is out of range, a structured coaching call will take place.
Change in Gestational Weight Gain at 36 Weeks Gestation | Baseline to 36 weeks gestation
  Body weight will be measured at each time point using Tanita MC-780U scale to assess gestational weight gain (GWG). Participants will use a BodyTrace scale linked to a secure monitoring system for weekly self-weighing monitored by health coaches. If weight is out of range, a structured coaching call will take place.
Change in Mean Arterial Pressure at 26 Weeks Gestation | Baseline to 26 Weeks Gestation
  Ambulatory monitoring negates the low sensitivity and specificity of clinical BP and could detect elevated BP, which is known to lead to pre-eclampsia. Data will be summarized to derive mean arterial pressure (MAP) by 24 hours and night time.
Change in Mean Arterial Pressure at 36 Weeks Gestation | Baseline to 36 Weeks Gestation
  Ambulatory monitoring negates the low sensitivity and specificity of clinical BP and could detect elevated BP, which is known to lead to pre-eclampsia. Data will be summarized to derive mean arterial pressure (MAP) by 24 hours and night time.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gamble, PhD, Principal Investigator — University of Mississippi Medical Center

IPD SHARING:
Plan to Share IPD: No